CLINICAL TRIAL: NCT06631560
Title: Hepatitis E Virus Infection in Oncological Patients - a Prospective Study in Rural Eastern Germany
Brief Title: Hepatitis E Virus Infection in Oncological Patients
Acronym: HepE-Onko-BB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Responsible Party: Principal Investigator, Isabel-Elena Haller, MD, Medizinische Hochschule Brandenburg Theodor Fontane
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HepE-Onko-BB
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Hepatitis E Infection; Hepatitis; Epidemic; Oncologic Disorders
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oncological disease (Experimental): Serum was taken from each patient before treatment initiation and during treatment follow-up. In addition, oncological participants completed a questionnaire consisting of eight questions focusing on quantitative aspects, to identify risk factors for HEV infection.
  Interventions: Diagnostic Test: ELISA testing
- Healthy controls (Experimental): Serum samples were analysed retrospectively using HEV ELISAs
  Interventions: Diagnostic Test: ELISA testing
- Control hospitalized due to SARS-CoV-2 infection (Experimental): Serum samples were analysed retrospectively using HEV ELISAs
  Interventions: Diagnostic Test: ELISA testing

INTERVENTIONS:
Diagnostic Test: ELISA testing — Diagnostic testing was performed by testing all serum samples using the HEV ELISA Wantai and Euroimmun kit.

SUMMARY:
The goal of this clinical trial is to investigate the prevalence of hepatitis E infection in oncological patients in a rural region of Germany. Consequently, we conducted prospective testing of blood samples from patients with haematological malignancies for evidence of HEV infection using two distinct anti-HEV IgG and IgM enzyme-linked immunosorbent assays (ELISAs). Serum was taken from each patient before treatment initiation and during treatment follow-up. Primary endpoint was determination of HEV seroprevalence. A healthy cohort was established alongside a cohort of patients who had been hospitalised due to a diagnosis of SARS-CoV-2 infection. In addition, oncological participants completed a questionnaire consisting of eight questions focusing on quantitative aspects, to identify risk factors for HEV infection.

ELIGIBILITY:
Inclusion Criteria:

* different hemato-oncological entities without age restriction

Exclusion Criteria:

* patients already receiving antineoplastic therapies
* not given written consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Anti HEV-IgM and IgG prevalences | In the oncological cohort, multiple samples were prospectively collected over a one-year period, commencing on 1 September 2020 and concluding at the end of October 2021. In the remaining two control samples, analysis was conducted retrospectively.
  Anti-HEV prevalences were determined in each arm with two different assays

SECONDARY OUTCOMES:
Identification of risk factors for HEV infection in oncological patients | The questionnaire was handed out at the beginning of the study
  Oncological participants completed a questionnaire consisting of eight questions focusing on quantitative aspects, to identify risk factors for HEV infection. Part of the questions were posed in a binary format, requiring a "yes" or "no" response. Additionally, we inquired as to the frequency with which risk factors such as pork are consumed. A multiple-choice format was employed, with the majority of questions comprising single-select multiple-choice options. To illustrate, the question for example enquired as to the frequency with which the patient consumed raw or undercooked pork products. The options ranged from "never" to "more than once a month".

CONTACTS AND LOCATIONS:
Overall Officials: Isabel-Elena Haller, Principal Investigator — Medical School (MHB) Theodor Fontane
Locations (1):
- Medical School (MHB) Theodor Fontane, Brandenburg, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: No